CLINICAL TRIAL: NCT05132374
Title: I-T CHILD: Building Babies' Brains With the Power of Healthy Relationships
Brief Title: The Infant- Toddler Climate of Healthy Interactions for Learning and Development (I-T CHILD)
Acronym: I-T CHILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Robinhood Foundation (Unknown); Adelphi University (Other); Docs for Tots (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000029873
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Child Development; Child Behavior; Social Skills; Infant Development
Keywords: low-income families; infants; toddlers; child care; home based; child care providers
MeSH Terms: conditions — Child Behavior; Social Skills

STUDY DESIGN:
Intervention Model Description: This study consists of the following main activities: (1) training and certification of early childhood mental health consultants from various agencies on the I-T CHILD Tool; (2) random assignment of child care providers into treatment (those receiving standard practice early childhood mental health consultation but enhanced with the I-T CHILD as a framework for consultation) and waitlist-control groups (no intervention until the end of the evaluation period); (3) provision of I-T CHILD resources to child care providers (user-friendly tips on how to strengthen their relationships with children and families); and (4) data collection (pre-test, post-test, 3-month follow-up).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Those receiving standard practice early childhood mental health consultation but enhanced with the I-T CHILD as a framework for consultation
  Interventions: Other: I-T CHILD
- Waitlist-control group (No Intervention): Those who receive no intervention until the end of the evaluation period)

INTERVENTIONS:
Other: I-T CHILD — This study will evaluate the I-T CHILD's application in early childhood mental health consultation services provided to family/group family child care programs
  Arms: Treatment Group

SUMMARY:
The purpose of the study is to train New York-based early childhood mental health consultants (ECMHCs) who will apply the Infant-Toddler Climate of Healthy Interactions for Learning and Development (I-T CHILD) tool as part of their standard practice. The study will evaluate I-T CHILD-informed early childhood mental health consultation in 100 New York State-licensed family day care and group family day care programs serving infants and toddlers in lower-income neighborhoods

DETAILED DESCRIPTION:
The overarching goal of the project is to provide New York City with the first strengths-based, equity-oriented, culturally responsive, and cost-efficient suite of measurement and caregiver-oriented tools designed to boost healthy brain development by both assessing and strengthening the quality of caregiver-infant/toddler relationships. The primary goal of the study is to evaluate the effectiveness of the I-T CHILD-informed ECMHC on the caregiver beliefs and teaching practices. The secondary goal is to assess whether changes in caregiver beliefs and teaching practices are associated with children's developmental outcomes.

This project is Phase 2 (RCT) of an earlier proof-of-concept of the I-T CHILD (Phase 1). Phase 2 evaluates the I-T CHILD's application in early childhood mental health consultation services provided to family/group family child care programs. Phase 2 consists of the following main activities: (1) training and certification of early childhood mental health consultants from various NY-based agencies on the I-T CHILD Tool; (2) random assignment of child care providers into treatment (those receiving standard practice early childhood mental health consultation but enhanced with the I-T CHILD as a framework for consultation) and waitlist-control groups (no intervention until the end of the evaluation period); (3) provision of I-T CHILD resources to child care providers (user-friendly tips on how to strengthen their relationships with children and families); and (4) data collection (pre-test, post-test, 3-month follow-up). Data to be collected will include caregiver self-report surveys, caregiver ratings of children, observations (live or remote, depending on COVID-19 guidelines), and amount of language used in the program using LENA technology. Additionally, qualitative data will be collected from consenting participants through phone (or Zoom) interviews, depending on participant preferences.

ELIGIBILITY:
Inclusion Criteria:

* Be operating a legal and licensed home-based child care program serving infants and toddlers

  o The program must serve at least one infant or one toddler, as the study and funding are centered around infants and toddlers.
* Agree to participate in a 3-month course of early childhood mental health consultation (ECMHC) provided by a trained ECMHC consultant beginning in about one month, if randomized to the treatment condition
* Agree to participate in data collection activities

  * Be able to respond to surveys either completed online via Yale Qualtrics surveys (home-based child care providers regularly submit licensing and child care subsidy forms online, so this should not be a challenge for legally-operating licensed child care providers), or by phone with a trained data collector.
  * Open to having blinded raters to observe the program.

Exclusion Criteria:

* Participants are excluded if they do not meet all of the inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the Framing Challenging Behaviors Questionnaire | Baseline, 4 Months and 8 Months
  a validated self-report questionnaire completed by child care providers that measures how they think about child misbehaviors. It includes 3 statements, on a 10 point scale continuum of two different thoughts or ideas regarding children's challenging behavior. Scores range between 1 to 10 (the mean score of the 3 statements). The continuum represents different ways of looking at children's misbehaviors, with higher scores representing a higher internal locus of control. It take 5 minutes or less to administer.
Change from baseline in Job Stress Inventory | Baseline, 4 Months and 8 Months
  a validated self-report questionnaire completed by child care providers that measures their level of child care provider job stress associated with their perceptions of job demands, job control, and job resources. It includes 22 statements, scored on a Likert 1-5 "How often..." ("Rarely/Never" to "Most of the Time"). The score range is 22- 110.The higher the score, the higher the perceived job stress level. It take 5 minutes or less to administer.
Change in Language Environment Analysis (LENA) | Baseline, 4 Months and 8 Months
  is a language analytic technology used for measuring the amount of language input received by infants and toddlers. The device records the sound environment within hearing range of the child throughout an entire day in the child care program through a vest. The LENA device is collected and connected to computer with LENA software installed. The LENA software processes the audio recordings into data metrics that include the child's exposure to verbal stimulation and number and complexity of child utterances. These metrices constitute the outcome variable in this area. More about LENA technology can be read here: https://www.lena.org/technology/. The child wears the vest for the entire day (8-12 hrs) while at the provider's home based childcare. The LENA system looks at adult word count (AWC); child vocalization count (CVC); and parent-child conversational turns (PCCTs) per hour.
Change from Baseline in CHILD for Home-Based Child Care Observation Tool | Baseline, 4 Months and 8 Months
  an observation measure of home-based child care environments for infants and toddlers adapted from a center-based child care version for preschoolers. It is completed by a trained observer during an approximately 2-hour observational period. Trainees achieve reliability in the course of a 3-day training program. The IT-CHILD is a comprehensive observational assessment of the mental health (or social and emotional) climate of early care and education settings. The measure consists of 28 easily observable items, scored on a 5-point anchored Likert scale ranging from -2 (very undermining) to +2 (very promoting). The score range is then -2 to +2. It takes approximately 2 hours of time to administer (20 minute observations followed by 10 minutes of interpretation and scoring for 4 sessions).
Change from Baseline in Infant-Toddler Risk of Expulsion assessment | Baseline, 4 Months and 8 Months
  a child care provider completed rating scale adapted from the validated Preschool Expulsion Risk Measure. The scale consists of 12 items rated on a 5-point Likert scale ("strongly disagree" to "strongly agree") that have been shown to accurately predict a child care providers intent to expel a child from the child care program. The score range is 1-4 (the mean score for the 12 statements), the higher the score, the higher the risk of expulsion).It take 5 minutes or less to administer.
Change from baseline in Devereux Early Childhood Assessment for Infants/Toddlers | Baseline, 4 Months and 8 Months
  is a validated measure of child development completed by the child care provider that measures an infant's or toddler's child overall development and social-emotional behaviors. It includes 33 statements (infant) or 36 statements (toddler), and is scored on a Likert scale of 0 to 4 ("Never" to "Very Frequently").Two standard scores are provided: percentile scores and T-scores. The T-scores are standard scores that have a set mean of 50 and a standard deviation of 10. T-scores on the DECA are categorized as follows: T-Scores of 60 and above indicate that the child has social and emotional "strengths," T-scores of 41-59 inclusive indicate that the child is showing a "typical" amount of positive behaviors related to social and emotional competence, and T-scores of 40 and below indicate that the child has a "need for instruction". It takes approximately 5- 10 minutes to administer.

SECONDARY OUTCOMES:
Change from baseline in Center for Epidemiological Studies Depression Scale | Baseline, 4 Months and 8 Months
  A standardized and validated self-report screening measure for depressive symptoms measured on Likert scale. The CED-D is one of the most widely used depression screeners for research purposes. The measure asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. It includes 10 statements, with a higher score indicating more reported depression. (two reverse scoring "I felt Happy" and "I felt hopeful about the future"). The possible range of the 10-item scale is 0 to 30, and a cut off score of ten or higher indicates the presence of significant depressive symptoms. It takes approximately 5 or less of time to administer.
Change from baseline in Adverse Childhood Experiences Survey | Baseline, 4 Months and 8 Months
  a standardized and validated self-report measure of events during a person's childhood that create stress and compromise health and mental health during their adult lives. 10 statements (parental divorce, homeless during childhood, etc.) are measured dichotomously (yes or no) based on whether or not they were experienced during childhood by the person completing the self-rating. The more 'yes' is answered, the more adverse childhood experience reported. People have an ACE score of 0 to 10. Each type of trauma counts as one, no matter how many times it occurs. It takes approximately 5 or less of time to administer.
Change from baseline in Brief Resilience Scale | Baseline, 4 Months and 8 Months
  a standardized and validated self-report measure of a person's resiliency or ability to bounce back from stress. It includes 6 statements, and is scored on a Likert scale (1-5, Strongly Disagree to Strongly Agree). To score, one adds the responses varying from 1-5 for all six items giving a range from 6-30. A higher score indicated a higher resiliency. It takes approximately 5 or less of time to administer.
Change from Baseline in Perceived Stress Scale | Baseline, 4 Months and 8 Monthss)
  is a standardized and validated self-report measure of the amount of stress a person is experiencing, using 10 items scored on a 5-point Likert scale 0-4 (Never to Very Often). The PSS is the most widely used scale for measuring the perception of stress. PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress. It takes approximately 5 or less of time to administer.
Change from Baseline in Positive and Negative Affect Scales | Baseline, 4 Months and 8 Months
  A validated self-report measure of overall positive and negative affect. It lists 20 adjectives describing positive (10 words) and negative feelings (10 words) (e.g., excited; ashamed) that a person generally feels on a five-point scale (very slightly to extremely). The scoring is the sum of positive feelings (10 words), and a sum of the negative feelings (10 words). Total scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect. It takes approximately 5 or less to administer.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Reyes, PhD, Principal Investigator — Yale University
Locations (1):
- Child care site name, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No